CLINICAL TRIAL: NCT00700440
Title: Phase II Study of Cetuximab Combined With Intensity Modulated Radiotherapy (IMRT) and Concurrent Chemotherapy of Cisplatin in Nasopharyngeal Carcinoma
Brief Title: Study of Cetuximab in Nasopharyngeal Carcinoma (NPC) With Chemoradiotherapy
Acronym: ENCORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sichuan Cancer Hospital and Research Institute (Other); Fujian Cancer Hospital (Other Government); Fudan University (Other); Cancer Hospital of Guizhou Province (Other); First Affiliated Hospital of Guangxi Medical University (Other); Central South University (Other)
Responsible Party: Departments of Radiation Oncology, Cancer Center, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR62202-770; PPRA-RTOG 0001
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2010-03-26 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2009-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Radiotherapy; chemotherapy; Drug Targeting; loco-regionally advanced nasopharyngeal carcinoma; Safety.; efficacy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): 400mg/m^2 intravenous infusion one week before radiotherapy, then 250mg/m^2 intravenous infusion weekly during radiotherapy
  Interventions: Drug: C225 (cetuximab)

INTERVENTIONS:
Drug: C225 (cetuximab) — one week before and then weekly during radiotherapy
  Other Names: Erbitux

SUMMARY:
This is an open, multicenter phase Ⅱ clinical trial on cetuximab (C225) combined with IMRT + concurrent chemotherapy of cisplatin in locoregionally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed prior to study entry
* Age between 18-69 years old
* Pathology approved to be nasopharyngeal carcinoma (types WHO Ⅱ-Ⅲ)
* Stage Ⅲ, Ⅳa, Ⅳb according to UICC (International Union Against Cancer) 2002 6th edition criteria
* Primary tumor measurable
* KPS score ≥80
* Expected life span ≥6 months
* Adequate bone marrow function: White Blood Cell≥4×109/L，Hemoglobin≥100g/L，Platelet≥100×109/L
* Adequate liver function: ALAT/ASAT<1.5 × upper limit of normal (ULN), bilirubin <1.5×ULN
* Adequate renal function: Creatinine Clearance < 1.5×ULN

Exclusion Criteria:

* Evidence of distant metastatic disease
* Surgical procedure of the primary tumor or lymph nodes (except diagnostic biopsy)
* Previous radiotherapy for the primary tumor or lymph nodes
* Previous exposure to epidermal growth factor-targeted therapy
* Prior chemotherapy or immunotherapy for the primary tumor
* Other previous malignancy within 5 years, except non-melanoma skin cancer or pre-invasive carcinoma of the cervix
* Any investigational agent prior to the 1st study medication
* Participation in another clinical study within the 30 days prior to Inclusion in this study.
* Peripheral neuropathy > grade 1
* Known grade 3 or 4 allergic reaction to any of the study treatment
* History of severe pulmonary or cardiac disease
* Creatinine Clearance < 30ml/min
* Know drug abuse / alcohol abuse
* Legal incapacity or limited legal capacity
* Active systemic infection
* Medical or psychiatric illness, which in the investigators' opinions, would not permit the subject to complete or fully and completely understand the risks and potential complications of the study
* Concurrent chronic systemic immune therapy or hormone therapy not indicated in the study protocol
* Pregnancy (confirmed by serum or urine β-HCG) or lactation period
* Severe intercurrent illness, e.g. uncontrolled hypertension, cardiac failure

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tai-xiang Lu, M.D., Principal Investigator — Departments of Radiation Oncology, Cancer Center, Sun Yat-sen University; Tong-yu Lin, M.D., PhD, Principal Investigator — Departments of Chemotherapy, Cancer Center, Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Sung FL, Poon TC, Hui EP, Ma BB, Liong E, To KF, Huang DP, Chan AT. Antitumor effect and enhancement of cytotoxic drug activity by cetuximab in nasopharyngeal carcinoma cells. In Vivo. 2005 Jan-Feb;19(1):237-45. PMID 15796181
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Kiss R, Salmon I, Pauwels O, Gras S, Danguy A, Etievant C, Pasteels JL, Martinez J. In vitro influence of gastrin, oestradiol and gonadotropin-releasing hormone on HCT-15 and LoVo human colorectal neoplastic cell proliferation. Eur J Cancer. 1991;27(10):1268-74. doi: 10.1016/0277-5379(91)90095-u. PMID 1835597
- [Background] Burtness B, Goldwasser MA, Flood W, Mattar B, Forastiere AA; Eastern Cooperative Oncology Group. Phase III randomized trial of cisplatin plus placebo compared with cisplatin plus cetuximab in metastatic/recurrent head and neck cancer: an Eastern Cooperative Oncology Group study. J Clin Oncol. 2005 Dec 1;23(34):8646-54. doi: 10.1200/JCO.2005.02.4646. PMID 16314626
- [Background] Curran D, Giralt J, Harari PM, Ang KK, Cohen RB, Kies MS, Jassem J, Baselga J, Rowinsky EK, Amellal N, Comte S, Bonner JA. Quality of life in head and neck cancer patients after treatment with high-dose radiotherapy alone or in combination with cetuximab. J Clin Oncol. 2007 Jun 1;25(16):2191-7. doi: 10.1200/JCO.2006.08.8005. PMID 17538164
- See also: Home Page of Chinese Anti-Cancer Association — http://www.caca.org.cn/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2008-7-1 ~ 2009-4-3
Period: Overall Study
Arm/Group | Cetuximab
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 0
Age Continuous [Median (Full Range); unit: Years] | 43 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 26
Region of Enrollment [Number; unit: participants]
  China | 100

OUTCOME MEASURES:

1. Primary Outcome: 3 Month Loco-regional Control After Cetuximab With Concurrent Chemoradiotherapy
Description: The response status (Complete Response + Partial Response) was evaluated according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria. Complete response was defined as disappearance of all target lesions, and Partial response was defined as at least a 30% reduction in the sum of the longest diameter of target lesions, taking as reference the baseline study.
  Adverse events of this combined modality treatment were graded according to CTCAE (Common Terminology Criteria for Adverse Events) v3.0 criteria.
Time Frame: 3 months
Measure: Number; unit: participants with loco-regional control
Arm/Group | Cetuximab
Number analyzed (Participants) | 100
participants with loco-regional control | 100

2. Secondary Outcome: 1,3,5 Year Loco-regional Control Rate, 1 Year Progression-free Survival and Metastasis-free Survival, 3 and 5 Year Overall Survival
Time Frame: 5 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less